CLINICAL TRIAL: NCT03839680
Title: Measuring Endoscopic ACTIvity in Patients Treated With VEDOlizumab for Ulcerative Colitis
Acronym: ACTIVEDO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2019/412
Record Dates: First submitted 2019-01-15; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis, endoscopic activity, mucosal healing, vedolizumab
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopy — The endoscopy procedure uses an endoscope to examine the interior of a hollow organ or cavity of the body.

SUMMARY:
Describe the proportion of patients with ulcerative colitis (UC) treated with vedolizumab (VDZ) who achieve mucosal healing at week 54 of treatment.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years,
* established diagnosis of ulcerative colitis for at least 3 months
* moderate to severe active ulcerative colitis with a Mayo endoscopic sub-score ≥ 1 before vedolizumab introduction
* patients receiving vedolizumab according to French drug labelling (previous exposure to anti-TNF, contraindicated or intolerant to anti-TNF),
* possibility of concomitant therapy including corticosteroids and immunosuppressors,
* patients naive to anti-integrin,
* no contraindication to proctosigmoidoscopy

Exclusion Criteria:

* age under 18 years
* ulcerative colitis not proven, Crohn's disease, or inderterminate colitis
* personal history of high-grade dysplasia or colorectal cancer
* surgery with ileo-anal anastomosis
* patients' refusal to participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients suffering from ulcerative colitis for who an endoscopic examen is performed
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-04-15 (Estimated); Study Completion 2019-04-15 (Estimated)

PRIMARY OUTCOMES:
Mucosal healing at defined by Mayo endoscopic sub-score ≤ 1 or UCEIS ≤ 1 | 54 weeks

SECONDARY OUTCOMES:
Mucosal healing at defined by Mayo endoscopic sub-score 0 or UCEIS 0 | 14 weeks
Mucosal healing at defined by Mayo endoscopic sub-score 0 or UCEIS 0 | 30 weeks
Mucosal healing at defined by Mayo endoscopic sub-score 0 or UCEIS 0 | 54 weeks
Endoscopic pattern of mucosal healing | 54 weeks

OTHER OUTCOMES:
Risk factors of mucosal healing | 14 weeks
  Risk factors will be assessed by consultation of patients medical record and reported on the spreedsheet for analysis:
  * Demographic data: age, gender, smoking habit
  * Characteristics of colitis: median duration of disease before starting VDZ, extension of disease according to the Montreal classification and severity at baseline (Mayo score/UCEIS)
  * Treatments:
  * Previous therapy used including number of TNF ɑ antagonist and reason for failure
  * Concomitant drugs: corticosteroids, immunosuppressors
  * Biologic tests with blood tests (Haemoglobin, CRP, albumin with dosage in patients 'referent laboratory or hospital laboratory priori to each infusion of VDZ) and fecal calprotectin, realized only in hospital laboratory due to repayment terms, from stool samples or aspiration during proctosigmoidoscopy.
Risk factors of mucosal healing | 30 weeks
  Risk factors will be assessed by consultation of patients medical record and reported on the spreedsheet for analysis:
  * Demographic data: age, gender, smoking habit
  * Characteristics of colitis: median duration of disease before starting VDZ, extension of disease according to the Montreal classification and severity at baseline (Mayo score/UCEIS)
  * Treatments:
  * Previous therapy used including number of TNF ɑ antagonist and reason for failure
  * Concomitant drugs: corticosteroids, immunosuppressors
  * Biologic tests with blood tests (Haemoglobin, CRP, albumin with dosage in patients 'referent laboratory or hospital laboratory priori to each infusion of VDZ) and fecal calprotectin, realized only in hospital laboratory due to repayment terms, from stool samples or aspiration during proctosigmoidoscopy.
Risk factors of mucosal healing | 54 weeks
  Risk factors will be assessed by consultation of patients medical record and reported on the spreedsheet for analysis:
  * Demographic data: age, gender, smoking habit
  * Characteristics of colitis: median duration of disease before starting VDZ, extension of disease according to the Montreal classification and severity at baseline (Mayo score/UCEIS)
  * Treatments:
  * Previous therapy used including number of TNF ɑ antagonist and reason for failure
  * Concomitant drugs: corticosteroids, immunosuppressors
  * Biologic tests with blood tests (Haemoglobin, CRP, albumin with dosage in patients 'referent laboratory or hospital laboratory priori to each infusion of VDZ) and fecal calprotectin, realized only in hospital laboratory due to repayment terms, from stool samples or aspiration during proctosigmoidoscopy.
Endoscopic response defined by a decrease in Mayo endoscopic sub-score ≥1 or decrease in UCEIS ≥ 2 points | 14 weeks
Endoscopic response defined by a decrease in Mayo endoscopic sub-score ≥1 or decrease in UCEIS ≥ 2 points | 30 weeks
Endoscopic response defined by a decrease in Mayo endoscopic sub-score ≥1 or decrease in UCEIS ≥ 2 points | 54 weeks
Clinical response defined by a decrease in the total Mayo score ≥ 3 points and ≥ 30 %, with a decrease in the sub score for rectal bleeding ≥ 1 or an absolute rectal-bleeding sub-score ≤ 1 | 14 weeks
Clinical response defined by a decrease in the total Mayo score ≥ 3 points and ≥ 30 %, with a decrease in the sub score for rectal bleeding ≥ 1 or an absolute rectal-bleeding sub-score ≤ 1 | 30 weeks
Clinical response defined by a decrease in the total Mayo score ≥ 3 points and ≥ 30 %, with a decrease in the sub score for rectal bleeding ≥ 1 or an absolute rectal-bleeding sub-score ≤ 1 | 54 weeks
Clinical remission defined by a total Mayo score ≤ 2 with no sub-score > 1 | 14 weeks
Clinical remission defined by a total Mayo score ≤ 2 with no sub-score > 1 | 30 weeks
Clinical remission defined by a total Mayo score ≤ 2 with no sub-score > 1 | 54 weeks
Histologic remission defined by a Nancy index score at 0 or 1 | 14 weeks
Histologic remission defined by a Nancy index score at 0 or 1 | 30 weeks
Histologic remission defined by a Nancy index score at 0 or 1 | 54 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU de Besançon, Besançon
  - CHU de Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - CHI de Haute-Saône, Vesoul

IPD SHARING:
Plan to Share IPD: No